CLINICAL TRIAL: NCT01240252
Title: Molecular Regulation of Muscle Glucose Metabolism in Man, Protocol 4
Brief Title: Insulin Receptor Substrate 1 (IRS-1) Regulation in Insulin Resistance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lawrence Mandarino, Professor, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10-003382; R01DK047936 (NIH)
Record Dates: First submitted 2010-09-29; First posted 2010-11-15 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Insulin; Insulin, Regular, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Type 2 Diabetes Mellitus Subjects (Experimental): Two hours after the start of deuterated glucose, subjects will receive human insulin (U100 Humulin) at a rate of 80 mU/m^2 surface area per minute one time over 4 hours.
  Interventions: Drug: Human insulin
- Overweight or Obese Subjects with Normal Glucose Tolerance (Experimental): Two hours after the start of deuterated glucose, subjects will receive human insulin (U100 Humulin) at a rate of 80 mU/m^2 surface area per minute one time over 4 hours.
  Interventions: Drug: Human insulin
- Non-Obese Control Subjects (Placebo Comparator): Two hours after the start of deuterated glucose, subjects will receive human insulin (U100 Humulin) at a rate of 80 mU/m^2 surface area per minute one time over 4 hours.
  Interventions: Drug: Human insulin

INTERVENTIONS:
Drug: Human insulin — U100 Humulin at a rate of 80 mU/m^2 surface area per minute one time over 4 hours
  Other Names: Humulin

SUMMARY:
The study is being conducted to find out why too much fat in your blood stream may cause insulin resistance in your muscles. Insulin is the hormone, produced normally by your body, which causes your blood sugar to return to normal after you eat.

DETAILED DESCRIPTION:
Insulin resistance in skeletal muscle is an early event in the pathogenesis of type 2 diabetes, obesity, and other conditions associated with the Metabolic Syndrome. The aim of this study is to determine the extent to which the inflammatory response to lipids is present in naturally occurring insulin resistance. We will test the hypothesis that skeletal muscle from insulin resistant volunteers is characterized by:

1. Increased concentrations of circulating proinflammatory cytokines without changes in cytokine expression in muscle.
2. Increased inflammatory response in muscle.
3. Increased infiltration of inflammatory cells into skeletal muscle.
4. Changes in expression of proteasome genes.

Forty five subjects will be studied in total. Three groups will be studied. One group will consist of 15 patients with type 2 diabetes mellitus The second group will consist of 15 age, gender, and body composition matched overweight or obese subjects (27 < BMI <36) with normal glucose tolerance. The third group will consist of 15 age and gender matched nonobese control subjects (BMI < 27).

There will be two visits in the study, a screening visit and the study visit. At visit 2 the subject will report to the study site having fasted since the night before, discuss the study and provide written consent, and provide a history and physical exam. Screening tests include a 12-lead resting EKG, complete blood chemistry and complete blood count (CBC), glycated hemoglobin (HbA1c), and a lipid profile. If the results of these tests show that the subject is eligible to participate in the study, a second visit will be scheduled. On the same day as the screening visit, the patient will have an oral glucose tolerance test.

Within 3 months of the screening visit, the subject will return after an overnight fast for a euglycemic clamp study and 2 muscle biopsies. Diabetic subjects will have oral medications discontinued for 3 days before study (metformin and thiazolidinedione treatment will be excluded). Patients taking insulin will have neutral protamine Hagedorn (NPH) discontinued the evening before study, and Glargine will be discontinued the morning and evening on the day before study. An antecubital catheter will be placed for infusion of substances. Deuterated glucose will be used to determine the rates of basal and insulin stimulated glucose uptake. A hand vein will be catheterized and placed in a heated box to arterialize venous blood for measurement of arterial glucose concentrations. One hour later, a percutaneous biopsy of the vastus lateralis muscle will be performed. Biopsy specimens (75-150 mg) will be frozen immediately in liquid nitrogen and stored in liquid nitrogen until they are processed. One hour after the muscle biopsy (two hours after the start of deuterated glucose), a primed-continuous (80 milliunits (mU)/(m^2 per min)) insulin infusion will be started and continued for 120 minutes to quantify the effects of insulin on glucose disposal. Throughout the insulin infusion, an infusion of 20% glucose will be adjusted to maintain euglycemia. Plasma glucose in the diabetics will be allowed to fall during the insulin infusion to euglycemia, where it will be maintained. A second muscle biopsy will be performed in the contralateral leg at the conclusion of the insulin infusion.

ELIGIBILITY:
Inclusion criteria:

* Age 30-65 y
* Healthy lean, obese, or known type 2 diabetic
* Body Mass Index (BMI) less than 36
* All nondiabetic subjects must have normal oral glucose tolerance
* Subjects must have the following laboratory values:

  1. Hematocrit ≥ 35 vol%
  2. Serum creatinine ≤ 1.6 mg/dl
  3. Aspartate aminotransferase (AST) (SGOT)< 2 times upper limit of normal
  4. Alanine aminotransferase (ALT) (SGPT)< 2 times upper limit of normal
  5. Alkaline phosphatase < 2 times upper limit of normal
  6. Triglycerides < 150 mg/dl
  7. Prothrombin time (PT) 11.7 -14.3 seconds
  8. Partial thromboplastin time 23.0-37.0 seconds

Exclusion criteria:

* No diseases known to affect glucose metabolism other than healthy type 2 diabetes
* Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded.
* Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
* Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>180, diastolic BP>105, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Proportion of insulin resistant patients with elevated serine/threonine phosphorylation of IRS-1 in muscle. | one month from date of volunteer study
  IRS-1 will be immunoprecipitated from percutaneous muscle biopsies, resolved by gel electrophoresis, digested with trypsin, and analyzed by high-performance liquid chromatography nanospray tandem mass spectrometry (MS/MS) analysis

SECONDARY OUTCOMES:
Quantitative assay of the ability of insulin to clear glucose from the blood in insulin resistant patients. | one month from date if volunteer study
  The glucose clamp gives a quantitative measure, in mass per unit body weight per minute, of the ability of insulin to cause glucose to disappear from the blood

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Mandarino, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States